CLINICAL TRIAL: NCT07167615
Title: CA-LINC Caring Connections Randomized Control Trial Study
Brief Title: Caring Connections Youth Suicide Prevention Care Coordination Study
Acronym: CA-LINC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Village Heartbeat, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-2167
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Suicide; Suicide Prevention; Suicide Ideation; Suicide Attempt
Keywords: youth; suicide prevention; care coordination; suicide intervention
MeSH Terms: conditions — Suicide; Suicide Prevention; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Caring Connections (Experimental): Caring Connections is a 90-day culturally adapted LINC intervention developed with and for youth. The Caring Connection intervention integrates engagement and follow-up strategies to assess/monitor suicide risk, facilitate service use referrals/linkages, develop/reﬁne safety plans, and create villages of care. The Caring Connections intervention incorporates culturally promotive factors, empowerment, and motivational strategies to support, enhance strengths, promote hope, improve family relationships, and reinforce caring messages. This consumer-, community-, and theory-driven care coordination intervention is designed to reduce suicide ideation and behavior (SIB) by improving service engagement and delivery standards. Caring Connections is implemented by Peer Support Specialists and Community Health Workers assigned to mental health "hubs" in Faith-Based Organizations (FBOs) to facilitate standardization and access to care.
  Interventions: Behavioral: Caring Connections
- Active Comparator: Treatment as Usual (Active Comparator): The treatment-as-usual arm includes care coordination services provided by Peer Support Specialists and Community Health Workers in the faith-based organization mental health hubs. This condition includes screening to determine youth suicide risk (high vs. low). Youth presenting with high risk are typically referred to an inpatient treatment facility. Youth presenting with low risk may be referred to a local outpatient provider. Mental health hub staff may attempt to follow up with families (typically not more than a one-time check-in) to ensure they are connected to the referral source. Following initial referrals, mental health hubs typically continue to provide crisis response and referral services to youth and caregivers as needed.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Caring Connections — Participants receive the Caring Connections intervention.
  Arms: Experimental: Caring Connections
Behavioral: Treatment as Usual (TAU) — Participants receive treatment as usual.
  Arms: Active Comparator: Treatment as Usual

SUMMARY:
The goal of this pilot randomized control trial (RCT) is to test the feasibility of Caring Connections, a Culturally Adapted Linking Individuals Needing Care (CA-LINC) suicide prevention care coordination intervention for high-risk suicidal youth. This consumer-, community-, and theory-driven care coordination intervention is designed to reduce suicide ideation and behavior (SIB) by improving service engagement. Connections is a 90-day intervention that integrates engagement and follow-up strategies to assess/monitor suicide risk, facilitate service use referrals/linkages, develop/reﬁne safety plans, and create villages of care. The intervention incorporates cultural promotive factors, empowerment, and motivational strategies aimed at supporting youth, enhancing strengths, promoting hope, improving family relationships, and reinforcing caring messages. Primary research questions include:

1. Is Caring Connections feasible to use for suicidal high-risk youth?
2. Does Caring Connections have the potential to reduce suicide ideation and behaviors among high-risk suicidal youth?

For the pilot RCT, 80 youth participants ages 13-19 who meet the inclusion criteria will be randomly assigned to one of two conditions: Caring Connections (n=40) or Treatment as Usual (n=40). Additionally, investigators will enroll 80 caregivers of youth meeting inclusion criteria and 20 Mental Healthcare, Healthcare Providers, Community Stakeholders, and/or Care Coordinators with experience working with suicidal youth. Researchers will compare those receiving Caring Connections with treatment as usual to see if suicidal ideation and behaviors, and engagement.

DETAILED DESCRIPTION:
Linking Individuals Needing Care (LINC) is a consumer- and theory-driven care coordination intervention designed to reduce suicidal ideations and behaviors by improving service engagement and delivery standards. However, LINC has not been culturally adapted to meet the specific needs of all youth and caregivers, nor has it been integrated with communities whose help-seeking behaviors are often facilitated through non-behavioral health supports. Caring Connections is a proposed adaptation of LINC to meet the specific needs of youth and families by incorporating input from communities whose help-seeking behaviors are often facilitated through non-behavioral health supports such as faith-based organizations. This study has the potential to improve service delivery standards and reduce suicide risk among youth.

Caring Connections is implemented by Peer Support Specialists and Community Health Workers assigned to mental health "hubs" in Faith-Based Organizations (FBOs) that facilitate standardization and access to care for youth/families regardless of religious affiliation. FBOs effectively mobilize communities to promote positive health behaviors.

The aims of this study are the following: (1) Assess stakeholder perceptions on the acceptability/appropriateness of the adapted intervention, (2) Assess provider and community stakeholder perceptions on the practicality and integration of implementing and sustaining Caring Connections using existing community resources/infrastructure, (3) Evaluate the feasibility of study procedures for screening, recruitment, and randomization, (4) Evaluate treatment adherence, fidelity, and study retention, (5) Examine effect size estimates for differences in primary outcomes (suicide ideation and behaviors (SIB) among youth randomly assigned to Caring Connections vs. Treatment as Usual (TAU), (6) Examine differences in potential change mechanisms (i.e., therapeutic alliance, service utilization, cultural humility, family relationships, engagement behaviors, and participation barriers) between Caring Connections and TAU.

All participants will participate in a care coordination intervention aimed at linking them to resources and decreasing their risk for suicide. For the randomized control trial, investigators will enroll 180 participants, including 80 youth ages 13-19 with recent suicidal ideation and behaviors (<90 days), 80 Caregivers of youth meeting inclusion criteria, and 20 Care Coordinators, Providers, or Community Stakeholders with experience working with youth. Upon consent, the measures/data collection will occur at baseline, 30, 90, and 180 days. Measures will be administered by IRB-compliant university research assistants (blinded to group assignment in the RCT).

This pilot will inform the feasibility, usability, and implementation of a novel care coordination approach aimed at addressing the lack of culturally responsive interventions for reducing youth suicide risk. Caring Connections will assess elements of feasibility (acceptability, practicality, integration) aimed to facilitate rapid uptake and sustainability within existing mental health "hubs'' embedded in FBOs. This study has potential for improving service delivery standards, reducing suicide risk among diverse youth populations,

ELIGIBILITY:
Inclusion Criteria:

Youth:

* 13 - 19 years old
* Current or recent history (<90 days) of suicide ideation, planning, or attempts or nonsuicidal self-injurious behaviors per youth or caregiver self-report or positive screen on the Patient Health Questionnaire Adolescent (PHQ-A), C-SSRS, or Ask Suicide-Screening Questions (ASQ).
* Able to fluently speak and read English
* Youth with a prior history of difficulty accessing services.
* Written assent to participate in the study (<18 years old)
* Written consent from a parent/legal guardian/caregiver to participate in the study (<18 years old)
* Written consent if the youth is ages 18-19

Parents/Legal Guardians/Caregivers:

* The primary caregiver of a youth who meets the above inclusion criteria for the study
* Over the age of 18
* Able to fluently speak and read English
* Without intellectual disabilities
* Provide written consent to participate

Mental Healthcare and/or Healthcare Providers and/or Community Stakeholders:

* Mental Health, behavioral health, substance use and/or health-related professionals who screen/assess for mental health and/or suicide risk or provide referrals, treatment, or follow-up care to youth with a prior history of difficulty accessing services in the surrounding treatment areas based on this risk or community stakeholder (i.e., faith-based leaders, agency directors, advocates, school administrators, hospital/crisis directors, topical experts, etc.).
* Over the age of 18
* Able to fluently speak and read English
* Without intellectual disabilities
* Provide written consent to participate

Care Coordinators:

* Care coordinators who screen/assess for mental health and/or suicide risk or provide referrals, treatment, or follow-up care to underserved youth in the surrounding treatment areas.
* Over the age of 18
* Able to fluently speak and read English
* Without intellectual disabilities

Exclusion Criteria:

Youth

* Youth at imminent suicide risk (reported verbally and/or indicated on C-SSRS)
* Youth who exhibit severe cognitive, language, or developmental delays
* Youth not meeting inclusion criteria

Parents/Legal Guardians/Caregivers:

* Not meeting the inclusion criteria listed above.

Mental Healthcare and/or Healthcare Providers and/or Community Stakeholders:

* Not meeting the inclusion criteria listed above.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Suicide Ideation Severity | Baseline, 30 days, 90 days, 180 days
  Investigators assess the suicide ideation severity using the Columbia-Suicide Severity Rating Scale (C-SSRS), a 6-item validated tool used to assess a person's risk for suicide. Assess suicidal ideation severity (5 items [yes/no]; scores range from 0 to 5, with higher scores indicating more severe suicidal ideation)
Reported Suicide Attempts | Baseline, 30 days, 90 days, 180 days
  Investigators will assess the presence of suicidal behaviors (yes/no) over the past month. Question #6 from the Columbia-Suicide Severity Rating Scale (C-SSRS) will be used which assesses a person's risk for suicide. A yes response indicates suicidal behaviors.

SECONDARY OUTCOMES:
Change in Treatment Acceptability | 30 days, 90 days
  The Treatment Evaluation Inventory Short Form (TEI-SF) is a 14-item, reliable, and valid measure that has been modified to assess the acceptability of CA-LINC. The total score ranges from 9 to 45, with higher scores indicating greater acceptability of the treatment.
Change in Therapeutic Alliance | 30 days, 90 days
  The Therapeutic Alliance Scales for Adolescents (TASA) is a reliable, valid 12-item scale slightly modified to assess the helping relationship between the youth/care coordinator. Scores range from 12 to 48, with higher scores indicating a stronger therapeutic alliance.
Change in Cultural Humility | 30 days, 90 days
  The Cultural Humility Scale (CHS) a reliable, valid 12-item scale to determine youth perceived cultural humility within the youth-care coordinator relationship. Scores range from 12 to 60, where higher scores indicate greater cultural humility.
Change in Family Relationships | Baseline, 30 days, 90 days, 180 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Family Relationship is a reliable, valid 47-item measure to assess youth's perceptions of family relationships. The measure provides a standardized T-score, where 50 represents the average for the general population, and scores are interpreted based on whether they are above (better family relationships) or below this average (worse family relationships).
Change in Engagement Behaviors | 30 days, 90 days
  The Engagement Behaviors Scale (EBS) is a 17-item measure, adapted from the Adolescent Alliance-Building Scale to assess helping behaviors of care coordinators. The scores range from 0 to 85, with higher scores indicating strong engagement behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Sonyia Richardson, Ph.D., Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication, provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become 9 to 36 months following publication and will remain available as long as the principal investigator remains actively working.
Access Criteria: See Plan Description section above for IRB or similar authorization prior to access. Once those criteria have been met, an interested investigator may contact the study PI by email (sonyia.richardson@unc.edu); the PI would arrange for deidentified data sharing in accordance with university policy.